CLINICAL TRIAL: NCT04425330
Title: The Effects of Physical Therapy Associated With Photobiomodulation on Functional Performance in Children With Low Lumbar and Sacral Myelomeningocele - A Randomized, Blinded Clinical Trial.
Brief Title: Effects of Physical Therapy Associated With Photobiomodulation on Myelomeningocele
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mielomeningocele
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Physical Therapy Modalities
Keywords: Meningomyelocele; Low-Level Light Therapy; Photobiomodulation; Neurological Rehabilitation
MeSH Terms: conditions — Meningomyelocele | interventions — phytobacteriomycin; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Participants will not know whether which group they are participating in, that is, treatment group or placebo with photobiomodulation.
  * The evaluator and who will perform the exercises will not know which group the participant is participating in relation to photobiomodulation.
  * A therapist who will not participate in assessments and physiotherapy sessions will perform the application of photobiomodulation.
  * The microtubes with the saliva samples will be marked with numbers corresponding to each participant, so the evaluator will not know which group the sample corresponds to. A therapist will be responsible for the assessment and electromyography scales.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physiotherapy exercises + PBM (Experimental): Physiotherapy exercises will be individualized and personalized for each child. It will take into account complaints and / or motor delay resulting from the injury. Circuit exercises will be performed involving muscle strengthening exercises, sensory stimulation and balance.
  For irradiation, the subjects will be positioned comfortably in prone position on the examination table. Four points will be irradiated above the injury level. The level of the lesion will be located by palpation. Four points will be irradiated above the injury level. The level of the lesion will be located by palpation. The irradiation will be with LED with a wavelength of 850 nm, energy per point of 25 J, 50 seconds per point and power of 200 mW.
  Treatment will be performed in 24 sessions 2 times a week
  Interventions: Other: physiotherapy exercises; Other: PBM
- physiotherapy exercises + SHAM PBM (Sham Comparator): Physiotherapy exercises will be individualized and personalized for each child. It will take into account complaints and / or motor delay resulting from the injury. Circuit exercises will be performed involving muscle strengthening exercises, sensory stimulation and balance.
  For irradiation, the subjects will be positioned comfortably in prone position on the examination table. Four points will be irradiated above the injury level. The level of the lesion will be located by palpation. The same LED device will be used in groups. However, in the placebo group (Sham), the device does not emit light.
  Treatment will be performed in 24 sessions 2 times a week
  Interventions: Other: physiotherapy exercises; Other: SHAM PBM

INTERVENTIONS:
Other: physiotherapy exercises — The evidence on the effectiveness of physical therapy in children with myelomeningocele is limited. The International Classification of Functionality, Disability and Health for Children and Youth is a useful tool to assist therapists in analyzing problems about the focus of the intervention. The evidence in physical therapy practice for individuals of all ages with neurological disorders, focuses on 5 Ps: prevention, prediction, participation, personalized and plasticity. Thus, neurological physiotherapists must perform the care with a focus on preventing the patient's disabilities, predicting the ideal response of an intervention, through measures of results of the movement system. In addition, it is of paramount importance that the goal of rehabilitation is that people with neurological disabilities are fully included and participate in life activities that are important to them and that their care is personalized. All of these measures facilitate the process of positive plasticity.
Other: PBM — Photobiomodulation occurs from the application of low intensity light such as low intensity laser and light emitting diode (LED). The therapeutic effectiveness of phototherapy is based on the absorption of photons by photoreceptors or chromophores. Studies on the experimental model of spinal cord injury have shown that both wavelengths have the potential to be an effective and non-invasive means of therapy, promoting axonal appearance, increased concentration of glial cells and nerve connections, in addition to functional and sensitive. The findings of a clinical trial involving individuals diagnosed with spinal cord injury demonstrate that PBM exerted positive effects on motor function, especially during isotonic contraction of stimulated muscles assessed by electromyography, and there was a recovery in sensory perception and muscle strength.
  Other Names: Low level laser therapy
  Arms: physiotherapy exercises + PBM
Other: SHAM PBM — SHAM PBM
  Arms: physiotherapy exercises + SHAM PBM

SUMMARY:
Myelomeningocele is a severe type of spina bifida, resulting from improper closure of the neural tube. This condition drastically affects the structures of the spinal cord, as a result the spinal cord, nerve roots and meninges are exposed during pregnancy resulting in deficiencies. The combination of these deficiencies results in an overall decrease in mobility and functional participation. There is little evidence about physical therapy interventions in this population. However, it is known that the International Classification of Functionality, Disability and Health for Children and Youth is a useful tool to assist therapists in analyzing problems and thinking about the focus of the intervention. The current literature demonstrates that resources such as low intensity light, also known as photobiomodulation as a therapeutic means, can be auxiliary means in the rehabilitation of neurological conditions, as studies show that photobiomoduction promotes sensory and motor recovery in the animal model of spinal cord injury . And a clinical trial showed that after photobiomodulation treatment combined with photobiomodulation, individuals with spinal cord injuries improved motor and sensory function. Therefore, the objective of the study is to evaluate the effects of physical therapy associated with photobiomodulation on functional performance in children with low and sacral lumbar myelomeningocele. Materials and methods: Participants will be recruited at the Integrated Health Clinic of University Nove de Julho. Those who meet the inclusion criteria will be randomized to two groups using a randomization site (randomization.com). Group 1 will be submitted to active PBM and physiotherapeutic exercises. Group 2 will be submitted to sham PBM and physiotherapeutic exercises. Irradiation will be carried out with LED at a wavelength of 850 nm, energy of 25 J per point, 50 seconds per point and a power of 200 mW. The same device will be used in the placebo group but will not emit light. Muscle activity will be assessed using a portable electromyograph (BTS Engineering) and the sit-to-stand task will be performed as a measure of functioning. Electrodes will be positioned on the lateral gastrocnemius, tibialis anterior and rectus femoris muscles. The Pediatric Evaluation of Disability Inventory will be used to assess the functional independence of the children. Quality of life will be assessed using the Child Health Questionnaire - Parent Form 50. Change in participation will be assessed using the Participation and Environment Measure for Children and Youth (PEM-CY). The sensory evaluation will be performed using the Semmes-Weinstein kit (AesthesioVR kit, California, EUA, DanMic Global). The protein expression of BDNF will be quantified from saliva samples using the ELISA technique. The data will be analyzed with the aid of GraphPad PRISM. The results of this study can contribute to a better understanding of the effectiveness of physiotherapy on the functionality and quality of life of children with myelomeningocele. In addition, FBM is a non-invasive treatment, and a fast procedure and can be a promising approach in the treatment

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of myelomeningocele on the lower lumbar and sacral level;
* able to perform the movement of sitting and standing with support

Exclusion Criteria:

* Cognitive impairment that compromises the ability to communicate
* Allergy to latex; neuromuscular scoliosis; subluxation or dislocation of the hip and knee;
* other disease of the central nervous system.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2020-11-03 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2022-02-03 (Estimated)

PRIMARY OUTCOMES:
Electromyography | 30 minutes
  Muscle activity will be assessed using a portable electromyography (BTS Engineering) synchronized to the BST EMG analyzer system. As a measure of functionality, the sit-to-stand task will be performed.
  The electrodes will be positioned on the muscles: lateral gastrocnemius, anterior tibialis and rectus femoris.
  For the assessment of the sit-to-stand the participant will be positioned in a chair with 90º flexion of the hip, knee, ankle and supported feet.
  An assessment will be carried out with the child sitting at rest. Afterwards, the child will be asked to stand up and remain in an upright position for 10 seconds. Afterwards the child will be asked to sit down. The repetition of the sit-to-stand task will be performed 3 times with an interval of 5 minutes.

SECONDARY OUTCOMES:
Sensory evaluation - monofilaments | 10 minutes
  The sensory evaluation will be performed using the Semmes-Weinstein kit (AesthesioVR kit, California, EUA, DanMic Global), which is a set of six nylon monofilaments of the same length that exert force on the specific area tested. Each monofilament has a different color and diameter: the kit contains 20 monofilaments, which exert different forces upon bending, with 20 target forces: 0.008 g;0.02 g, 0.04 g, 0.07 g, 0.16 g, 0.40 g, 0.60 g, 1.0 g, 1.4 g, 2.0 g, 4.0 g, 6.0 g, 8.0 g, 10 g, 15 g, 26 g, 60 g, 100 g, 180 g, and 300 g.). The test will be performed on the following dermatomes: L1, L2, L4, L5, S1, S2.
Assessment of functional skills | 10 minutes
  To assess the functional independence of children, the Pediatric Evaluation of Disability Inventory (PEDI) will be used. This child assessment tool assesses functional performance, in terms of capabilities (functional skills) and performance of what the child actually does in response to the environment (the amount of caregiver assistance needed to perform daily tasks) in three domains: self-care, mobility and social function. This inventory was translated into Portuguese and culturally adapted to take into account Brazilian socio-cultural specificities.
Quality of life assessment | 10 minutes
  The quality of life will be assessed through the Child Health Questionnaire - Parent Report 50 (Child Health Questionnaire - Parent Form 50 - CHQ-PF50), which is a useful tool, since it allows to evaluate this aspect from the parents' perspective.
BDNF evaluation | 5 minutes
  Protein expression of BDNF will be quantified from saliva samples using the ELISA technique. DELUXE HUMAN commercial kit (BioLegend®) will be used. The analysis will be according to the manufacturer's instructions. The optical density of the samples will be measured on the spectrophotometer at 450 nm.
Participation and Environment Measure | 40 minutes
  The PEM-CY is a parent-report instrument that examines participation and environment factors that affect the participation of children across three settings: home, school, and community.

REFERENCES:
- [Derived] Silva T, Queiroz JR, Turcio KHL, Tobelem DDC, Araujo TR, Coutinho KSL, Chavantes MC, Horliana ACRT, Deana AM, Silva DFTD, Castelo PM, Fernandes KPS, Motta LJ, Mesquita-Ferrari RA, Kalil Bussadori S. Effect of photobiomodulation combined with physical therapy on functional performance in children with myelomeningocele: A protocol randomized clinical blind study. PLoS One. 2021 Oct 6;16(10):e0253963. doi: 10.1371/journal.pone.0253963. eCollection 2021. PMID 34613973